CLINICAL TRIAL: NCT06710197
Title: IL-1 Inhibition for Patients With Early Stage Triple Negative and ER-low Breast Cancer: a Window-of-opportunity Study
Brief Title: IL-1 Inhibition in Early TNBC
Acronym: OZM-034
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WOO-11-2023
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Early Stage Triple Negative ER Low Breast Cancer
Keywords: WOO
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: This study will examine changes in the tumor microenvironment (TME) induced by 14 days of pre-operative IL-1-inhibiting therapy among patients with early breast cancer (including TNBC and ER-low positive [1-9%]). Key immune biomarkers (TILs, TAMs, NK cells, IL-1β and inflammasome component expression) will be evaluated at baseline and following 14 days of IL-1 antagonist therapy (Anakinra) using paired tissue specimens. A total of 50 patients will be recruited across 2-5 institutions, randomized 4:1 to treatment (n=40) versus control (n=10).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Anakinra SC injection 100mg daily x 14 days
  Interventions: Drug: Anakinra (Kineret®)
- Group 2 (No Intervention): Patients will receive standard of care treatment

INTERVENTIONS:
Drug: Anakinra (Kineret®) — 100 mg/daily subcutaneously
  Arms: Group 1

SUMMARY:
This study will examine changes in the tumor microenvironment (TME) induced by 14 days of pre-operative IL-1-inhibiting therapy among patients with early breast cancer (including TNBC and ER-low positive). Key immune biomarkers (TILs, TAMs, NK cells, IL1[beta] and inflammasome component expression) will be evaluated at baseline and following 14 days of IL-1 antagonist therapy (Anakinra) using paired tissue specimens.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in this study, patients must fulfill all the following criteria:

  1. Age > 18 years
  2. Histologically confirmed non-metastatic invasive adenocarcinoma of the breast meeting one of the following criteria:

     i. Clinical stage T1a/b N0 TNBC ii. Clinical stage T1a/b N0 ER-low (1-9%)
  3. Not planned for neoadjuvant chemotherapy

Exclusion Criteria:

Patients who satisfy any of the following exclusion criteria are NOT eligible for this study.

1. Male Gender
2. HER2 positive breast cancer
3. Second primary cancer
4. Multifocal early breast cancer
5. Pre-existing inflammatory arthritis
6. Pregnancy or lactating.
7. Platelets ≤ 100x109/L. ANC ≤ 1.5 x109/L. Hemoglobin ≤ 80 g/L
8. ECOG≥2
9. Clinically significant bacterial, fungal, parasitic or viral infection, which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
10. Known active hepatitis A, B, C or who are HIV-positive or who are at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Prior test results obtained as part of standard of care that confirm a subject is immune and not at risk for reactivation (i.e., hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility and tests do not need to be repeated. Subjects with prior positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
11. Primary immunodeficiency such as X-linked agammaglobulinemia or common variable immunodeficiency.
12. Active and inactive ('latent') tuberculosis infection or suspicion of active tuberculosis. If no suspicion of active tuberculosis, testing is not required.
13. Use of glucocorticoids above the equivalent of 10 mg of prednisone daily within 4 weeks prior to treatment with Anakinra.
14. Major surgery within 4 weeks prior to treatment.
15. History of malignancy in the past 3 years except for treated, early-stage squamous or basal cell carcinoma of the skin or carcinoma-in-situ of the cervix.
16. History or current diagnosis of uncontrolled or significant cardiac disease, including any of the following: a. myocardial infarction within last 6 months. b. uncontrolled congestive heart failure. c. unstable angina within last 6 months. d. exertional angina. e. clinically significant (symptomatic) cardiac arrhythmias (e.g., bradyarrhythmia, sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker).
17. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
18. Presence of moderate or severe renal function impairment (estimated creatinine clearance <60 mL/min/1.73m2).
19. Patients with mild, moderate, or severe hepatic impairment or inadequate liver function defined by any of direct bilirubin, alanine amino transferase (ALT), or aspartate aminotransferase (AST)>2.5 x upper limit of normal (ULN). Patients with Child-Pugh score >5 are also excluded.
20. Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 30 days of screening or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
21. Significant concurrent, uncontrolled medical condition which, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
22. Known hypersensitivity to E-coli derived proteins, Anakinra or any component of the product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In this study, we will enroll women with early TNBC or ER low (1-9%) breast cancer with lesions that clinically measure up to 1cm in size (T1a/T1b), or lesions that are between 1 and <2cm (T1c) with no clinical evidence of lymph node involvement who are not planned for neoadjuvant chemotherapy.
Enrollment: 50 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To determine the changes in the breast cancer TME in paired patient samples (core biopsy and surgical specimen) before and after 14 days of treatment with the IL-1 receptor antagonist, Anakinra. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network-Princess Margaret Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided